CLINICAL TRIAL: NCT02153489
Title: A Pilot, Double-blind, Placebo-controlled, 2-period Crossover Study to Assess the Effect of Aclidinium Bromide 400 μg Bid on COPD Symptoms and Sleep Quality After 3 Weeks of Treatment in Patients With Stable Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Double-blind, Placebo-controlled, Crossover Study to Assess the Effect of Aclidinium Bromide 400 μg Bid on COPD Symptoms and Sleep Quality After 3 Weeks of Treatment in Patients With Stable Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M/34273/47; 2013-003373-10 (EudraCT Number)
Record Dates: First submitted 2014-05-05; First posted 2014-06-03 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aclidinium bromide (Experimental): Aclidinium bromide 400 μg administered via oral inhalation (Genuair® dry powder inhaler) one inhalation twice daily (12 hours apart, morning and evening).
  Interventions: Drug: Aclidinium bromide
- Placebo (Placebo Comparator): Placebo administered via oral inhalation (Genuair® dry powder inhaler) one inhalation twice daily (12 hours apart, morning and evening).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium bromide
  Other Names: Eklira®
  Arms: Aclidinium bromide
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of aclidinium bromide compared with placebo in improving dilatation of the airways (bronchodilation), symptoms of chronic obstructive pulmonary disease (COPD), sleep quality and physical activity after 3 weeks of treatment with aclidinium bromide 400 μg administered twice daily in patients with stable moderate-and-severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or non-pregnant, non-lactating female aged ≥40 years. Women of childbearing potential will follow specific study requirements (negative serum pregnancy test at the Screening Visit and are using, over the last two months before the Screening Visit, at least one medically approved and highly effective method of birth control
* Current or ex-cigarette smoker (patients who quit smoking more than 6 months prior to the Screening Visit), with a smoking history of at least 10 pack-years.
* Patients with a clinical diagnosis of chronic obstructive pulmonary disease (COPD) according to GOLD guidelines 2013, with a post bronchodilator FEV1 <80%, and FEV1 ≥ 40% at Screening Visit
* Patients must be able to perform repeatable pulmonary function testing for FEV1 according to American Thoracic Society [ATS]/European Respiratory Society [ERS] 2005 criteria at Screening Visit
* Patients who are eligible and able to participate in the study and who consents to do so in writing after the purpose and nature of the investigation have been explained

Exclusion Criteria:

* History or current diagnosis of asthma
* Patients with moderate to severe sleep apnoea assessed at screening
* Patients who develop a respiratory tract infection or COPD exacerbation within 6 weeks (or 3 months if hospitalisation was required) before the Screening Visit (Visit 1) or during the run-in period
* Clinically significant respiratory conditions
* Patients with Type I or uncontrolled Type II diabetes, uncontrolled hypo-or hyperthyroidism, hypokalaemia, or hyperadrenergic state, uncontrolled or untreated hypertension
* Patients who may need to start a pulmonary rehabilitation program during the study and/or patients who started/finished it within 3 months prior to the Screening Visit
* Use of long-term oxygen therapy (15 hours/day)
* Patients who does not maintain regular day/night, waking/sleeping cycles including night shift workers
* Clinically significant cardiovascular conditions
* QTc >470 milliseconds in the manual ECG reading performed at Screening Visit
* Patients with clinically relevant abnormalities in the opinion of the investigator at the Screening Visit (Visit 1) in the results of the clinical laboratory tests, ECG parameters or in the physical examination)
* Patients with a history of hypersensitivity reaction to inhaled anticholinergics, long and short acting β2-agonists, sympathomimetic amines, or inhaled medication or any component there of (including report of paradoxical bronchospasm)
* Patients with known narrow-angle glaucoma, symptomatic bladder neck obstruction, acute urinary retention, or patients with symptomatic non-stable prostatic hypertrophy
* Patients with known non-controlled history of human immunodeficiency virus (HIV) infection and/or active hepatitis
* History of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years other than basal or squamous cell skin cancer
* Patients with any other serious or uncontrolled physical or mental dysfunction, or moderate-to-severe depression, as confirmed by Beck Depression Inventory (BDI-II) total score >28.
* Patients with a history (within 2 years prior to the Screening Visit) of drug and/or alcohol abuse that may prevent study compliance based on investigator judgment
* Patients unlikely to be cooperative or that can't comply with the study procedures.
* Patients treated with any investigational drug within 30 days (or 6 half-lives, whichever is longer) prior to the Screening Visit
* Patients who intends to use any concomitant medication not permitted by this protocol or who have not undergone the required stabilization periods for prohibited medication
* Any other conditions that, in the investigator's opinion, might indicate the patient to be unsuitable for the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ribera, PhD, Study Director — AstraZeneca Barcelona
Locations (2):
- Germany (2):
  - Pulmonary Research Institute at the Lung Clinic Grosshansdorf, Großhansdorf
  - Pneumologische Lehrklinik der Universitätsmedizin Göttingen, Immenhausen

REFERENCES:
- [Derived] Magnussen H, Arzt M, Andreas S, Plate T, Ribera A, Seoane B, Watz H, Kirsten AM. Aclidinium bromide improves symptoms and sleep quality in COPD: a pilot study. Eur Respir J. 2017 Jun 22;49(6):1700485. doi: 10.1183/13993003.00485-2017. Print 2017 Jun. No abstract available. PMID 28642315

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by 3 investigators at 3 sites in Germany. The first patient was screened in April 2014 and the last patient visit was in June 2015
Pre-assignment Details: All patients who met the study entry criteria and completed the screening assessments and the 7-day run-in period were randomized. Nine (9/39) subjects were not randomized due to screening failure (primarily for non-fulfillment of inclusion/exclusion criteria)
Groups:
- Sequence A: Aclidinium 400 μg - Placebo
- Sequence B: Placebo - Aclidinium 400 μg
Period: Period 1
Arm/Group | Sequence A | Sequence B
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence A | Sequence B
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All patients participating in the crossover study
Arm/Group | Overall Study
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Normalized Forced Expiratory Volume in One Second (FEV1) AUC0-24hr
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 11, 12, 12.5, 13, 14, 15, 16, 19, 22, 23, and 24 hours at Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: L/sec*hr
Groups:
- Aclidinium: Aclidinium 400 μg BID
- Placebo: Placebo BID
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
L/sec*hr | 0.0953 (0.0381) | -0.0429 (0.0381)

2. Other Pre Specified Outcome: Change From Baseline in Morning Trough FEV1
Time Frame: Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: Liters/sec
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Liters/sec | 0.1128 (0.0395) | -0.0106 (0.0395)

3. Other Pre Specified Outcome: Change From Baseline in Peak FEV1
Time Frame: Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: Liters/sec
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Liters/sec | 0.1605 (0.0391) | -0.0149 (0.0391)

4. Other Pre Specified Outcome: Change From Baseline in Normalized FEV1 AUC0-12hr
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 11 and 12 hours at Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: L/sec*hr
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
L/sec*hr | 0.1394 (0.0406) | -0.0100 (0.0406)

5. Other Pre Specified Outcome: Change From Baseline in Normalized FEV1 AUC12-24hr
Time Frame: 12, 12.5, 13, 14, 15, 16, 19, 22, 23, and 24 hours at Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: L/sec*hr
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
L/sec*hr | 0.0513 (0.0369) | -0.0758 (0.0369)

6. Other Pre Specified Outcome: Change From Baseline in the Average Rating of Overall Early Morning COPD Symptom Severity
Description: Night-time and early-morning symptoms were recorded every morning using the Early-Morning Symptoms of COPD Instrument [EMSCI] and the Night-time Symptoms of COPD Instrument [NiSCI]. Scores ranged from 0 (no symptoms) to 4 (very severe symptoms). The questionnaires also evaluated nocturnal awakenings and limitation of early-morning activities (scores ranged from 0 [no limitation] to 4 [a very great deal]). Symptoms assessed over 24 weeks included change from baseline in the severity of night-time and early-morning cough, wheezing, shortness of breath and difficulty bringing up phlegm, overall night-time and early-morning symptom severity, number of nocturnal awakenings and limitation of early-morning activities due to COPD symptoms
Time Frame: Week 3 of treatment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Score on a scale | -0.07 (0.575) | 0.09 (0.476)

7. Other Pre Specified Outcome: Change From Baseline in the Average Rating of Overall Evening COPD Symptom Severity
Description: The evening symptoms questionnaire was filled out after the second medication administration of the day and before bedtime. Scores ranged from 0 (no symptoms) to 4 (very severe symptoms). Symptoms assessed over 24 weeks included change from baseline in the severity of evening cough, wheezing, shortness of breath and tightness of the chest, chest congestion, difficulty bringing up phlegm, overall evening symptom severity, and limitation of evening activities due to COPD symptoms
Time Frame: Week 3 of treatment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Score on a scale | -0.15 (0.661) | 0.11 (0.559)

8. Other Pre Specified Outcome: Change From Baseline in the Average Rating of Overall Night-time COPD Symptom Severity
Description: as for outcome 6
Time Frame: Week 3 of treatment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Score on a scale | -0.14 (0.612) | -0.03 (0.526)

9. Other Pre Specified Outcome: Change From Baseline in the Average Rating of COPD Symptoms Limiting Early Morning Activities
Description: as for outcome 6
Time Frame: Week 3 of treatment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Score on a scale | -0.02 (0.457) | 0.16 (0.430)

10. Other Pre Specified Outcome: Change From Baseline in the Average Rating of COPD Symptoms Limiting Evening Activities
Description: as for outcome 7
Time Frame: Week 3 of treatment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Score on a scale | -0.18 (0.488) | 0.03 (0.450)

11. Other Pre Specified Outcome: Change From Baseline in Apnea-hypopnea Index (AHI) Per Hour of Total Sleep Time
Description: The Apnea Hypopnea Index (AHI) is used to indicate the severity of obstructive sleep apnea. The AHI is the number of apneas or hypopneas recorded during the study per hour of sleep
Time Frame: Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: Events/hr
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Events/hr | 0.4767 (0.4478) | 0.7700 (0.4478)

12. Other Pre Specified Outcome: Change From Baseline in Oxygen Desaturation Index (ODI) Per Hour of Total Sleep Time
Description: The oxygen desaturation index (ODI) is the number of times per hour of sleep that the blood's oxygen level drop by a certain degree from baseline. In this study, any event with a 4% decrease in blood oxygen levels counted towards the total
Time Frame: Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: Events/hr
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Events/hr | -0.3033 (0.9754) | 2.2400 (0.9754)

13. Other Pre Specified Outcome: Change From Baseline in Proportion of Sleep Stage REM as a Percentage of Total Sleep Time
Time Frame: Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: Percentage of total sleep time
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Percentage of total sleep time | 1.4100 (0.9851) | -1.1167 (0.9851)

14. Other Pre Specified Outcome: Change From Baseline in Sleep Efficiency
Description: Sleep efficiency is calculated as the total sleep time as a proportion of total time in bed
Time Frame: Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: Percentage of total time in bed
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Percentage of total time in bed | 1.0000 (2.4046) | -2.5500 (2.4046)

15. Other Pre Specified Outcome: Change From Baseline in Total Sleep Time
Time Frame: Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Minutes | 6.9200 (11.5802) | -11.8500 (11.5802)

16. Other Pre Specified Outcome: Change From Baseline in Duration of at Least Moderate Activity
Description: Moderate activity was defined as any physical activity >3 metabolic equivalents
Time Frame: Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Minutes | 9.4460 (6.7081) | -8.5943 (6.5879)

17. Other Pre Specified Outcome: Change From Baseline in Number of Steps Per Day
Time Frame: Week 3 of treatment
Measure: Least Squares Mean (Standard Error); unit: Number of steps per day
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 30 | 30
Number of steps per day | 268.5891 (326.3649) | 22.2652 (320.6754)

ADVERSE EVENTS:
Time Frame: Up to 30 days after last study drug administration
Arm/Group | Aclidinium | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium (N=30) | Placebo (N=30)
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the Investigator will be subject to mutual agreement between the investigator and sponsor.